CLINICAL TRIAL: NCT03678545
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy of Dupilumab (Anti-IL4a) in Subjects With Eosinophilic Gastritis
Brief Title: Dupilumab in Eosinophilic Gastritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0798; U54AI117804 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-09-19 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-03

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Gastroenteritis
MeSH Terms: conditions — Eosinophilic enteropathy | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either drug or placebo, followed by an open label extension
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Active Comparator)
  Interventions: Drug: Dupilumab (blinded)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (blinded)

INTERVENTIONS:
Drug: Dupilumab (blinded) — Subcutaneous injection every two weeks as follows: 600 mg initial dose, and 300 mg subsequent doses for a total of 6 injections.
  Arms: Dupilumab
Drug: Placebo (blinded) — Placebo is matched to the active drug (dupilumab), and is given in the same manner: a subcutaneous injection every two weeks for a total of 6 injections.
  Arms: Placebo

SUMMARY:
40 participants with Eosinophilic Gastritis 12-70 years of age will be randomly assigned with dupilumab or placebo subcutaneous injections every two weeks for a total of 12 weeks. Study subjects who complete the 12-week treatment phase, may continue into an open label extension study, where dupilumab will be administered every two weeks for a total of 24 weeks.

DETAILED DESCRIPTION:
This is a phase 2, multi-center, randomized, double-blind, placebo-controlled trial testing the efficacy of dupilumab vs. placebo in EG. Qualifying subjects will be randomized 1:1 to either study drug (dupilumab) or placebo, and will receive 600 mg once followed by 300 mg doses every two weeks of study treatment for a total of 6 injections. After the 6th injection subjects may continue into an open-label treatment phase in which dupilumab will be administered every two weeks for a total of 24 weeks.

Approximately 14 sites associated with the Consortium of Eosinophilic Gastrointestinal Disease Researchers (CEGIR) will take part in the study.

The primary objective of this study is to assess the efficacy of repeat subcutaneous (SC) doses of dupilumab, compared with placebo, to reduce eosinophilic inflammation in the gastrointestinal tract of patients with EG.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent guardian must be able to understand and provide informed consent and/or assent.
2. Willing and able to comply with study visits and activities
3. Age ≥ 12 and < 71 years at study enrollment
4. Histologically active EG at time of screening, with a peak gastric count of ≥ 30 eos/hpf in at least 5 hpfs in the gastric antrum and/or body.
5. History (by patient report) of moderate to severe EG symptoms
6. Stable medical management of EG.
7. Willing to maintain current dietary regimen throughout the course of the study. Diet must have been stable for 8 weeks prior to baseline endoscopy.
8. If have asthma and/or any other chronic allergic conditions they must be willing to maintain their pretrial medications until the end of study. Medication dose can be increased if there is a deterioration in the condition.
9. Score on Asthma Control Test (ACTTM) ≥ 20

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Current active H. pylori infection.
3. Systemic gastrointestinal disorders such as Crohn's disease, inflammatory bowel disease, or Celiac disease.
4. Known or suspected active colitis in the Principal Investigator's opinion or by biopsy.
5. Hypereosinophilic syndrome.
6. History of cancer
7. Current or recent use of biological agents.
8. Leukocyte count has not returned to the relevant lower limit of normal after discontinuing cell depleting biological agents.
9. Current or recent use of any investigational drug.
10. Current use of systemic steroids with daily dose > 10 mg for any reason or steroid burst for > 3 days within 1 month of screening.
11. Prior exposure to dupilumab.
12. History of anaphylaxis to any biologic therapy.
13. Current pregnancy or breastfeeding.
14. Ocular disorder.
15. Individuals who have required use of a systemic corticosteroid for asthma.
16. Received live vaccine 30 days prior to screening or planning on receiving a live vaccine during the time period that he/she is participating in the study.
17. Any esophageal stricture unable to be passed with a standard, diagnostic upper endoscope.
18. History of bleeding disorders or esophageal varices.
19. Active parasitic infection.
20. History of alcohol or drug abuse within 6 months prior to screening.
21. Participant or his/her immediate family is a member of the investigational team.
22. Planned or anticipated major surgical procedure during the study.
23. Initiation, discontinuation or addition of allergens to subcutaneous immunotherapy (SCIT) within 12 months prior to screening.
24. Treatment with sublingual immunotherapy (SLIT) within 6 months prior to screening.
25. Treatment with oral immunotherapy (OIT) within 6 months prior to screening.
26. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals or antifungals within 2 weeks before the baseline visit
27. Known or suspected immunodeficiency disorder, including human immunodeficiency disorder (HIV).
28. Planned or anticipated use of any prohibited medications and procedures during the study.
29. Initiation, discontinuation or change in the dosage regimen of the following Proton pump inhibitors (PPIs) Leukotriene inhibitors Nasal and/or inhaled corticosteroids
30. Women of childbearing potential who are unwilling to practice highly effective contraception.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rothenberg, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (12):
- United States (12):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - Northwestern Medicine Digestive Health Center, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
data will be collected from 14 different sites and kept in a secure electronic database supported by the NIH: Rare Diseases Data Management and Coordinating Center. Information such as test results, eligibility and patient reported outcomes can be accessed by authorized personnel from each site. staff from each site will only have access to the data collect by that site. The main site, CCHMC, will have full access to all data collected from all sites.

REFERENCES:
- [Derived] Sia T, Bacchus L, Tanaka R, Khuda R, Mallik S, Leung J. Dupilumab Can Induce Remission of Eosinophilic Gastritis and Duodenitis: A Retrospective Case Series. Clin Transl Gastroenterol. 2024 Jan 1;15(1):e00646. doi: 10.14309/ctg.0000000000000646. PMID 37753954

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (blinded): Placebo is matched to the active drug (dupilumab), and is given in the same manner: a subcutaneous injection every two weeks for a total of 6 injections.
  Open Label extension Placebo group to be treated with dupilumab.
Period: Double Blinded Phase
Arm/Group | Dupilumab | Placebo
Started | 21 | 20
Completed | 21 | 19
Not Completed | 0 | 1
Period: Open Label Extension
Arm/Group | Dupilumab | Placebo
Started | 21 | 19
Completed | 20 | 17
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dupilumab | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants] — Years
  Participants
    <=18 years | 5 | 5 | 10
    Between 18 and 65 years | 16 | 15 | 31
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (12.9) | 30.7 (14.0) | 30.4 (13.45)
Age, Continuous [Mean (Full Range); unit: years] | 30.3 [12 to 57] | 30.7 [12 to 59] | 30.4 [12 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Relative Change of Peak Eosinophil Counts in the Stomach
Description: We will determine the Relative change from baseline of the peak eosinophil counts in the 5 most eosinophil dense HPFs in the gastric antrum and/or body between drug vs placebo at 12 weeks will be the primary measurement endpoint.
Time Frame: 12 weeks after randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Eosinophil per HPF (EOS/HPF)
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 21 | 19
Eosinophil per HPF (EOS/HPF) | -50.28 [-66.20 to -34.37] | -3.54 [-20.27 to 13.19]

ADVERSE EVENTS:
Time Frame: From informed consent to 4 weeks after the end of the 12-week double-blind, approximately 20 weeks on average, followed by open-label treatment phase of 24 weeks. approximately a total of 44 weeks.
Groups:
- Experimental Phase - Dupilumab: Dupilumab (blinded): Subcutaneous injection every two weeks as follows: 600 mg initial dose, and 300 mg subsequent doses for a total of 6 injections.
- Experimental Phase - Placebo: Placebo (blinded): Placebo is matched to the active drug (dupilumab), and is given in the same manner: a subcutaneous injection every two weeks for a total of 6 injections.
- Open Label Phase - Dupilumab: Post experimental phase, all participants were offered an open-label extension.
Arm/Group | Experimental Phase - Dupilumab | Experimental Phase - Placebo | Open Label Phase - Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/40
Other Adverse Events (participants affected / at risk) | 19/21 | 18/20 | 37/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Phase - Dupilumab (N=21) | Experimental Phase - Placebo (N=20) | Open Label Phase - Dupilumab (N=40)
Eosinophilia (Blood and lymphatic system disorders) | 6 (10) | 5 (7) | 8 (21)
Cardiovascular events - Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain/Swelling (Eye disorders) | 0 (0) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection reaction (General disorders) | 12 (30) | 4 (5) | 19 (59) — Non-cardiac chest pain, Malaise, injection site reaction
Allergic reaction (Immune system disorders) | 1 (2) | 0 (0) | 1 (1)
Infections (Infections and infestations) | 6 (8) | 9 (12) | 15 (25)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) — bruising and non-study related flesh wounds
Low iron (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal irritations (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 6 (6) — muscular pain and joint pain
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cold like symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 3 (4) | 4 (8) — sore throat, nasal congestion, cough, wheezing
Rashes (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 5 (6)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infraction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Watery eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
EOG symptoms worsened (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Priapism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03678545/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03678545/SAP_001.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03678545/ICF_002.pdf